CLINICAL TRIAL: NCT02856438
Title: An Expanded Access Program for Elotuzumab in Combination With Lenalidomide Plus Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma in Japan
Brief Title: Early Patient Access Treatment Use Protocol CA204-220
Status: No longer available | Type: Expanded Access
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: CA204-220
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — Specified dose on specified days
  Other Names: BMS-901608
Drug: Lenalidomide — Specified dose on specified days
Drug: Dexamethasone — Specified dose on specified days

SUMMARY:
The objective of this expanded access program is to provide treatment with elotuzumab in combination with lenalidomide and dexamethasone for patients with relapsed or refractory multiple myeloma at Japanese sites where licensed physicians determine clinical need.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria

* Men and women 20 years and older.
* Active, relapsed or refractory multiple myeloma by International Myeloma Working Group (IMWG) criteria as assessed by the treating physician and have received at least 1 prior line of multiple myeloma therapy.
* Progression from a most recent line of therapy.
* Prior lenalidomide exposure is permitted only if they fulfill all of the following:.

  i) Were not refractory to prior lenalidomide, defined as no progression while receiving lenalidomide (induction dose) or within 60 days of last dose of lenalidomide. Patients progressing on lenalidomide maintenance dose are eligible for enrollment.

ii) Patient did not discontinue lenalidomide due to a Grade ≥ 3 related AE.

Exclusion Criteria

* All Adverse Events of any prior chemotherapy, surgery, or radiotherapy not resolved to NCI CTCAE (v. 3.0) Grade ≤ 2.
* Significant cardiac disease as determined by the treating physician including cardiac amyloidosis.
* HIV infection or active hepatitis A, B, or C.
* Any medical conditions that, in the attending physician's opinion, would impose excessive risk to the patient.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- Japan (3):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Shibukawa-shi, Gunma
  - Local Institution, Osaka, Osaka

REFERENCES:
- See also: EAP Investigator Requests — http://www.bms.com/clinical_trials/investigator_sponsored_research/Pages/expanded-access-program.aspx
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm